CLINICAL TRIAL: NCT06813495
Title: Prevention of Injuries Among Nurses and Nursing Aides Using Eastern Principles Acceptance and Commitment Therapy: Clinical Trial and Dissemination Research
Brief Title: Eastern Principles Acceptance and Commitment Therapy For Injury Prevention Among Nurses and Nursing Aides
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bowling Green State University (Other)
Collaborators: Ohio Bureau of Workers Compensation (Unknown)
Responsible Party: Principal Investigator, Willliam H. O'Brien, Professor at Department of Psychology, Bowling Green State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10011559
Record Dates: First submitted 2024-10-09; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Well-Being, Psychological; Work Injury; Musculoskeletal Pain; High Frequency Heart Rate Variability; Burnout; Mindfulness; Self-Compassion; Acceptance and Commitment Therapy; Heart Rate Variability
MeSH Terms: conditions — Psychological Well-Being; Musculoskeletal Pain; Burnout, Psychological | interventions — Nurses

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eastern Principles Acceptance and Commitment Therapy for Nurss and Nursing Aids (EPACT NNA) (Active Comparator): The EPACT intervention is designed to promote psychological flexibility (Hayes, et al., 2006), compassion, a recognition of impermanence, common humanity, and non-self-attachment. Psychological flexibility has six core processes: acceptance, cognitive defusion, present moment awareness, self-as-context, values, committed action. The EPACT NNA intervention will be group-based with 5-10 participants per group. The group-based format has been shown to be an effective delivery method for NNAs (O'Brien, et al., 2019b). The EPACT NNA protocol is comprised of two 2.5-hour sessions spaced one week apart.
  Interventions: Behavioral: Eastern Principles Acceptance and Commitment Therapy for Nurses and Nursing Aids (EPACT NNA)
- Acceptance and Commitment Therapy for Nurses and Nursing Aids (ACT NNA) (Active Comparator): The ACT NNA intervention has been previously tested for NNAs. It contains the six core processes identified above and omits the added EPACT components of acceptance of suffering, common humanity, impermanence, self- and other-compassion, and non-self- attachment. It will be delivered in a similar group-based format of 5-10 participants in three 2.5 - hour sessions.
  Interventions: Behavioral: Acceptance and Commitment Therapy for Nurses and Nursing Aids (ACT NNA)
- Control Group (No Intervention): Control group participants will complete measures at the same time points as the EPACT NNA and ACT NNA groups. We opted to use a no-treatment control group to allow for measurement of the durability of treatment gains across a 3-month follow-up period without an expectation for treatment.

INTERVENTIONS:
Behavioral: Eastern Principles Acceptance and Commitment Therapy for Nurses and Nursing Aids (EPACT NNA) — The EPACT intervention will be group-based with 5-10 participants per group. The group-based format has been shown to be an effective delivery method for NNAs (O'Brien, et al., 2019b). The EPACT protocol is comprised of two 2.5-hour sessions spaced one week apart.
  Arms: Eastern Principles Acceptance and Commitment Therapy for Nurss and Nursing Aids (EPACT NNA)
Behavioral: Acceptance and Commitment Therapy for Nurses and Nursing Aids (ACT NNA) — The ACT for NNA intervention has been previously tested for NNAs. It contains only the six core processes identified above and omits the added EPACT components of acceptance of suffering, common humanity, impermanence, self- and other-compassion, and non-self-attachment. It will be delivered in a similar group-based format of 5-10 participants in two 2.5 -hour sessions.
  Arms: Acceptance and Commitment Therapy for Nurses and Nursing Aids (ACT NNA)

SUMMARY:
This clinical trial will evaluate the effectivness of an Eastern Principles Acceptance and Commitment Therapy intervention (EPACT) relative to an estabished traditional Western-based Acceptance and Commitment Therapy intervention (ACT) and a no treatment control group. The participants for the study will be nurses and nursing aides (NNAs) who work in long-term care settings in the USA and Thailand. The primary dependent variables are work-related injuries, work stress and burnout, wellbeing, musculoskeletal symptoms, time off from work due to injury. High frequency heart rate variability will also be investigated as a predictor of responsiveness to the interventions.

The study has three primary aims:

1. To compare the EPACT NNA intervention to an established traditional Western ACT NNA intervention and a no-treatment control group.
2. To identify predictors of ACT NNA and EPACT NNA responsiveness to the interventions and injury likelihood across time.
3. To assess EPACT NNA's feasibility and effectiveness across cultures.

USA participants working in Ohio will be randomly assigned to one of three groups: EPACT NNA (n = 80), ACT NNA (n = 80), or a no treatment control group (n = 80). All participants will participate in an assessment session where study questnnaires are completed and a baseline high frequency HRV measurement is collected. Subsequent to the assessment, the EPACT NNA and ACT NNA participants will attend two 2.5 hour sessions spaced one week apart. The control group will have no further in-person meetings with the researchers. One-month after completing the intervention (4 weeks after the baseline assessment) a follow-up survey will be sent to participants for the first follow-up. Three months after baseline, the second follow-up survey will be sent to participants.

The surveys assess demographic characteristics, organizational variables, work-related injuries, work stress, and well-being.

A second RCT study will be conducted in Thailand comparing EPACT NNA (n = 40) to a no-treatment control group (n = 40) among nurses and nursing aides working in healthcare settings. The same outcome measures and procedures will be used.

This research aims to develop a culturally-informed, evidence-based intervention that integrates both Western and Eastern mindfulness principles to address the high rates of work-related injuries among NNAs.

DETAILED DESCRIPTION:
Nurses and nursing aides (NNAs) in healthcare settings are a diverse, vulnerable group who experience high rates of psychological and physical injuries. Addressing work-related injuries among NNAs is crucial for health, social, economic, and humanitarian reasons.

Research has shown that mindfulness predicts injuries among Ohio NNAs. A mindfulness-based intervention (Acceptance and Commitment Therapy, ACT) was effective in reducing injury-related absences and improving psychological wellbeing. However, Western mindfulness interventions may miss critical Eastern elements. It has been argued that Western "McMindfulness" interventions lack essential Eastern teachings, potentially reducing effectiveness, especially for healthcare workers.

Acceptance of suffering, self-compassion/loving-kindness, acceptance of impermanence, letting go of stress, nonself-attachment, and a common humanity are Eastern elements missing in Western mindfulness interventions. In collaboration with Thai mindfulness scholars, the researchers developed the Eastern Perspectives-added Acceptance and Commitment Therapy (EPACT NNA) for NNAs, integrating Eastern theories into an existing ACT protocol for NNAs. We hypothesize that EPACT NNA will more effectively reduce psychological and physical injuries, improve psychophysiological well-being, and shorten recovery times compared to conventional Western interventions or no treatment.

Specific Aim 1: Conduct a randomized clinical trial to evaluate EPACT NNA's effectiveness against traditional ACT for NNAs and a no-treatment control group. Outcome variables include: Psychological distress, injuries, well-being, work stress, burnout, compassion, psychological flexibility, and behavioral outcomes.

Specific Aim 2: Predict the responsiveness to EPACT NNA and the likelihood of psychological and physical injuries using on baseline measures of psychological and physiological functioning.

Specific Aim 3: Evaluate the feasibility and effectiveness of EPACT NNA in healthcare settings in Ohio and Thailand.

These aims align with NIH and Ohio BWC goals for preventing musculoskeletal and related injuries, integrating health and wellness into occupational safety, and improving mental health among workers. Additionally, this project acknowledges the Eastern origins of mindfulness practices.

The EPACT intervention will be group-based with 5-10 participants per group. The EPACT protocol is comprised of two 2.5-hour sessions spaced one week apart. The ACT for NNA intervention has been previously tested for NNAs. It contains only the six core processes identified above and omits the added EPACT components of acceptance of suffering, common humanity, impermanence, self- and other-compassion, and non-self- attachment. It will be delivered in a similar group-based format of 5-10 participants in two 2.5-hour sessions.

Control group participants will complete measures at the same time points as the EPACT and ACT groups. The researchers opted to use a no-treatment control group to allow for measurement of the durability of treatment gains across a 3-month follow-up period without an expectation for treatment.

All NNAs agreeing to participate will be asked to complete the informed consent and the pretreatment measures. The first EPACT and ACT for NNAs sessions will follow the pretreatment assessment. The control group will have not further in-person contact with researchers but will receive text and email messages. The following week, the ACT NNA and EPACT NNA participants will attend the second session. Exposure to violence, injury, musculoskeletal symptoms, burnout, mindfulness, and compassion measures will be completed at pretreatment, post-treatment, and three-months follow-up. Participants will complete these measures online. Heart rate variability will be assessed at pretreatment.

ELIGIBILITY:
Inclusion Criteria:

* USA: Employed as a nurse or nursing aide in a long-term care facility within a 120 mile radius of Bowling Green, Ohio.
* Thailand: Employed as a nurse or nursing aide in Chiang Mai, Thailand or Krung Thep Bangkok), Thailand.
* At least 18 years of age.
* Able to attend scheduled assessment and intervention appointments.

Exclusion Criteria:

• There are no a-priori exclusion criteria. However, if a participant reports significant psychological distress or a diagnosable mental health condition at the baseline assessment, they will be referred for an alternative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Organizational and Work Characteristics Associated with Injury | Measured at baseline (pretreatment), 1 month, and 3 months
  The Risk for Nursing Aide Injury Inventory (RNAII) contains 6 items measuring demographic variables, 9 items measuring job characteristics (e.g., tenure, hours per week, hours per shift, etc.) and 120 items assessing individual and organizational characteristics (e.g., staffing, space, training, physical environment characteristics, organizational constraints, incivility, family-work conflict, lifting device availability, organizational safety climate, supervisor relationships, and worker respect).
Exposure to Violence | Measured at baseline (pretreatment), 1 month, and 3 months
  The Workplace Violence Tool is used to measure exposure to assault and abuse of NNAs. The workplace violence tool consists of 7 items that assess the occurrence of: (a) threat of assault, (b) emotional abuse (e.g., hurtful remarks), (c) physical abuse (e.g., spit, kick, punch), (d) verbal sexual harassment, (e) sexual assault (e.g., touching, groping), and (f) forced sexual intercourse. Bostrom et al. (2011) modified the original measure to include information about the source of assault or abuse (resident, family member, coworker, other).
Work-related Injuries and Days Missed Due to Injury | Measured at baseline, 1 month, and 3 months
  The National Nursing Assistant Survey (NNAS) will be used to measure NNA injuries. The NNAS was developed by the Centers for Disease Control (Squillace, et al., 2007). The NNAS contains 6 items assessing musculoskeletal injuries, strains and muscle pulls, bites, scratches, wounds, cuts, bruising, and other types of injuries. Additionally, the NNAS measures the type of injury, cause of injury, days unable to work due to injury, and restricted activity due to injury.
Musculoskeletal Symptoms | Measured at baseline (pretreatment), 1 month, and 3 months
  Musculoskeletal symptoms will be measured a scale developed by Kuorinka et al. (1987). This scale asks participants how often they experienced any of 9 common musculoskeletal complaints, on a scale from "never" to "very often." The 9 complaints included in this scale adequately represent the musculoskeletal symptoms identified in our prior research with nursing aides (O'Brien et al., 2019a).
Burnout | Measured at baseline (pretreatment), 1 month, and 3 months
  Copenhagen Burnout Inventory (Kristensen, et al., 2005) will be used to measure burnout. The 18 items on the inventory form three subscales: personal burnout, work-related burnout, and client-related burnout. The scale has demonstrated strong reliability, consistency, and validity in prior research investigations.
Acceptance, present-moment awareness, self-as-context, defusion, values, and committed action | Measured at baseline (pretreatment), 1 month, and 3 months
  The Multidimensional Psychological Flexibility Inventory (MPFI) is a 60-item measure that was developed by Rolffs et al., (2018). The MPFI includes six subscales that measure psychological flexibility: acceptance, defusion, values, committed action, present-moment-awareness, self-as-context, and experiential avoidance. Six other subscales represent psychological inflexibility: experiential avoidance, fusion, lack of values, inaction, noncontact with the present moment, and self-as-content.
Self-compassion and other compassion | Measured at baseline (pretreatment), 1 month, and 3 months
  The Self-Compassion Scale (SCS) is a 26 item self-report measure that was developed by Neff (2003) to measure the extent to which a person may report a perspective towards the suffering of self that reflects kindness versus judgement, common humanity versus isolation, and mindfulness versus overidentification.
  The SCS yields 6 subscales: Self-Kindness, Common Humanity, Mindfulness, Self-Judgement, Isolation, and Over-Identified. The Compassion scale (CS) is a 16-item inventory measuring compassion for others. It has four subscales: kindness, common humanity, mindfulness, and lessened indifference.
Ubiquity of suffering, impermanence, common humanity, nonattachment to self. | Measured at baseline (pretreatment), 1 month, and 3 months
  The Mindfulness Insight Scale (MIS) is a 16-item measure that assesses the three characteristics of existence (inevitability of suffering, impermanence, and nonself-attachment/interconnectedness) from an Eastern and Buddhist perspective. Each item (e.g., "No living creature can escape suffering," "With or without noticing, change constantly occurs to everything," "I try not to get caught up in "Who I am.") is rated from 1 (very untrue) to 5 (very true).
High Frequency Heart Rate Variability (HF-HRV) | Measured at baseline (pretreatment), 1 month, and 3 months
  Resting HF-HRV levels will be collected from participants at their worksites. The resting HF-HRV will be recorded across a 10-minute interval while the participants are seated comfortably in a private room at each site. ECG data will be collected with a Biopac MP150 interfaced with Biopac Acqknowledge 4.3 software. ECG electrodes will be attached to participants using a lead II configuration. The ECG signal will be sampled at a rate of 1000Hz, which exceeds the minimum recommended sampling rate of 500Hz (Allen, et al., 2007). Once recorded, ECG signals will be replayed and visually inspected by researchers to detect and remove artifacts. The cleaned ECG data will then be analyzed using Kubios software (Tarvainen, et al., 2014).

CONTACTS AND LOCATIONS:
Locations (1):
- Bowling Green State University, Bowling Green, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Background] Ahola K, Salminen S, Toppinen-Tanner S, Koskinen A, Vaananen A. Occupational burnout and severe injuries: an eight-year prospective cohort study among Finnish forest industry workers. J Occup Health. 2013;55(6):450-7. doi: 10.1539/joh.13-0021-oa. Epub 2013 Oct 26. PMID 24162145
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Bernal D, Campos-Serna J, Tobias A, Vargas-Prada S, Benavides FG, Serra C. Work-related psychosocial risk factors and musculoskeletal disorders in hospital nurses and nursing aides: a systematic review and meta-analysis. Int J Nurs Stud. 2015 Feb;52(2):635-48. doi: 10.1016/j.ijnurstu.2014.11.003. Epub 2014 Nov 15. PMID 25480459
- [Background] Blignault I, Ponzio V, Rong Y, Eisenbruch M. A qualitative study of barriers to mental health services utilisation among migrants from mainland China in south-east Sydney. Int J Soc Psychiatry. 2008 Mar;54(2):180-90. doi: 10.1177/0020764007085872. PMID 18488410
- [Background] Bohlmeijer E, ten Klooster PM, Fledderus M, Veehof M, Baer R. Psychometric properties of the five facet mindfulness questionnaire in depressed adults and development of a short form. Assessment. 2011 Sep;18(3):308-20. doi: 10.1177/1073191111408231. Epub 2011 May 17. PMID 21586480
- [Background] Bos EH, Krol B, Van Der Star A, Groothoff JW. The effects of occupational interventions on reduction of musculoskeletal symptoms in the nursing profession. Ergonomics. 2006 Jun 10;49(7):706-23. doi: 10.1080/00140130600578005. PMID 16720530
- [Background] Bostrom AM, Squires JE, Mitchell A, Sales AE, Estabrooks CA. Workplace aggression experienced by frontline staff in dementia care. J Clin Nurs. 2012 May;21(9-10):1453-65. doi: 10.1111/j.1365-2702.2011.03924.x. Epub 2011 Dec 12. PMID 22151034
- [Background] Brown, R. L., & Moloney, M. E. (2018). Intersectionality, Work, and Well-Being: The Effects of Gender and Disability. Gender & Society, 33(1), 94-122. doi.org/10.1177/0891243218800636
- [Background] Burton A, Burgess C, Dean S, Koutsopoulou GZ, Hugh-Jones S. How Effective are Mindfulness-Based Interventions for Reducing Stress Among Healthcare Professionals? A Systematic Review and Meta-Analysis. Stress Health. 2017 Feb;33(1):3-13. doi: 10.1002/smi.2673. Epub 2016 Feb 25. PMID 26916333
- [Background] Chang YJ, Kwon YC, Lee WJ, Do YR, Seok LK, Kim HT, Park SR, Hong YS, Chung IJ, Yun YH. Burdens, needs and satisfaction of terminal cancer patients and their caregivers. Asian Pac J Cancer Prev. 2013;14(1):209-16. doi: 10.7314/apjcp.2013.14.1.209. PMID 23534725
- [Background] Chen Y, Yang X, Wang L, Zhang X. A randomized controlled trial of the effects of brief mindfulness meditation on anxiety symptoms and systolic blood pressure in Chinese nursing students. Nurse Educ Today. 2013 Oct;33(10):1166-72. doi: 10.1016/j.nedt.2012.11.014. Epub 2012 Dec 20. PMID 23260618
- [Background] Cohen, A., & Golan, R. (2007). Predicting absenteeism and turnover intentions by past absenteeism and work attitudes. Career Development International, 12(5), 416-432. doi.org/10.1108/13620430710773745
- [Background] Cohen-Katz J, Wiley SD, Capuano T, Baker DM, Kimmel S, Shapiro S. The effects of mindfulness-based stress reduction on nurse stress and burnout, Part II: A quantitative and qualitative study. Holist Nurs Pract. 2005 Jan-Feb;19(1):26-35. doi: 10.1097/00004650-200501000-00008. PMID 15736727
- [Background] Crenshaw, K. (1989) Demarginalizing the Intersection of Race and Sex: A Black Feminist Critique of Antidiscrimination Doctrine, Feminist Theory and Antiracist Politics, University of Chicago Legal Forum: Vol. 1989: Iss. 1, Article 8.
- [Background] Dantas EM, Sant'Anna ML, Andreao RV, Goncalves CP, Morra EA, Baldo MP, Rodrigues SL, Mill JG. Spectral analysis of heart rate variability with the autoregressive method: what model order to choose? Comput Biol Med. 2012 Feb;42(2):164-70. doi: 10.1016/j.compbiomed.2011.11.004. Epub 2011 Dec 2. PMID 22136799
- [Background] Dekker SW. Reconstructing human contributions to accidents: the new view on error and performance. J Safety Res. 2002 Fall;33(3):371-85. doi: 10.1016/s0022-4375(02)00032-4. PMID 12404999
- [Background] Duncan SM, Hyndman K, Estabrooks CA, Hesketh K, Humphrey CK, Wong JS, Acorn S, Giovannetti P. Nurses' experience of violence in Alberta and British Columbia hospitals. Can J Nurs Res. 2001 Mar;32(4):57-78. PMID 11928302
- [Background] Elliott, R., & Wexler, M. M. (1994). Measuring the impact of sessions in process- experiential therapy of depression: The Session Impacts Scale. Journal of Counseling Psychology, 41(2), 166. doi/10.1037/0022-0167.41.2.166
- [Background] Ghawadra SF, Abdullah KL, Choo WY, Phang CK. Mindfulness-based stress reduction for psychological distress among nurses: A systematic review. J Clin Nurs. 2019 Nov;28(21-22):3747-3758. doi: 10.1111/jocn.14987. Epub 2019 Jul 22. PMID 31267619
- [Background] Gloster, A. T., Walder, N., Levin, M. E., Twohig, M. P., & Karekla, M. (2020). The empirical status of acceptance and commitment therapy: A review of meta-analyses. Journal of Contextual Behavioral Science, 18, 181-192. doi.org/10.1016/j.jcbs.2020.09.009
- [Background] Goldberg, D. (1978). Manual of the general health questionnaire. Windsor, Ontario, Canada: National Foundation for Educational Research.
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hayes SC, Hofmann SG, Stanton CE. Process-based functional analysis can help behavioral science step up to novel challenges: COVID - 19 as an example. J Contextual Behav Sci. 2020 Oct;18:128-145. doi: 10.1016/j.jcbs.2020.08.009. Epub 2020 Aug 25. PMID 32864323
- [Background] Hayes SC, Hofmann SG. The third wave of cognitive behavioral therapy and the rise of process-based care. World Psychiatry. 2017 Oct;16(3):245-246. doi: 10.1002/wps.20442. No abstract available. PMID 28941087
- [Background] Haynes, S. N., O'Brien, W. H., & Keawe'aimoku Kaholokula, J. (2011). Behavioral assessment and functional analysis. Hoboken, NJ: Wiley.
- [Background] Henrich J, Heine SJ, Norenzayan A. The weirdest people in the world? Behav Brain Sci. 2010 Jun;33(2-3):61-83; discussion 83-135. doi: 10.1017/S0140525X0999152X. Epub 2010 Jun 15. PMID 20550733
- [Background] Horan, K. A., Moeller, M. T., Singh, R. S., Wasson, R., O'Brien, W. H., Matthews, R. A., Jex, S. M., & Barratt, C. L. (2018). Supervisor support for stress management and intervention process. International Journal of Workplace Health Management, 11(4), 260-272. doi.org/10.1108/ijwhm-12-2017-0113
- [Background] Jarvelin-Pasanen S, Sinikallio S, Tarvainen MP. Heart rate variability and occupational stress-systematic review. Ind Health. 2018 Nov 21;56(6):500-511. doi: 10.2486/indhealth.2017-0190. Epub 2018 Jun 16. PMID 29910218
- [Background] Jarukasemthawee, S., Halford, W. K., & McLean, J. P. (2019). When East meets West: A randomized controlled trial and pre- to postprogram evaluation replication of the effects of insight-based mindfulness on psychological well-being. Journal of Psychotherapy Integration, 29(3), 307-323. doi.org/10.1037/int0000179
- [Background] Kabat-Zinn, J. (1990). Full catastrophe living: Using the wisdom of your body and mind to face stress, pain and illness. New York: Delacorte
- [Background] Khatutsky, G., Wiener, J., Anderson, W., & Porell, F. (2012). Work-related injuries among certified nursing assistants in nursing homes. RTI Press publication No. RR-0017- 1204. Research Triangle Park, NC: RTI Press.
- [Background] Klein A, Taieb O, Xavier S, Baubet T, Reyre A. The benefits of mindfulness-based interventions on burnout among health professionals: A systematic review. Explore (NY). 2020 Jan-Feb;16(1):35-43. doi: 10.1016/j.explore.2019.09.002. Epub 2019 Oct 3. PMID 31727578
- [Background] Koeter MW. Validity of the GHQ and SCL anxiety and depression scales: a comparative study. J Affect Disord. 1992 Apr;24(4):271-9. doi: 10.1016/0165-0327(92)90112-j. PMID 1578083
- [Background] Kristensen, T. S., Borritz, M., Villadsen, E., & Christensen, K. B. (2005). The Copenhagen Burnout Inventory: A new tool for the assessment of burnout. Work & Stress, 19(3), 192-207. doi/10.1080/02678370500297720
- [Background] Kuorinka I, Jonsson B, Kilbom A, Vinterberg H, Biering-Sorensen F, Andersson G, Jorgensen K. Standardised Nordic questionnaires for the analysis of musculoskeletal symptoms. Appl Ergon. 1987 Sep;18(3):233-7. doi: 10.1016/0003-6870(87)90010-x. PMID 15676628
- [Background] Liu CH, Meeuwesen L, van Wesel F, Ingleby D. Why do ethnic Chinese in the Netherlands underutilize mental health care services? Evidence from a qualitative study. Transcult Psychiatry. 2015 Jun;52(3):331-52. doi: 10.1177/1363461514557887. Epub 2014 Dec 2. PMID 25468826
- [Background] Mackenzie CS, Poulin PA, Seidman-Carlson R. A brief mindfulness-based stress reduction intervention for nurses and nurse aides. Appl Nurs Res. 2006 May;19(2):105-9. doi: 10.1016/j.apnr.2005.08.002. PMID 16728295
- [Background] McGinn KL, Oh E. Gender, social class, and women's employment. Curr Opin Psychol. 2017 Dec;18:84-88. doi: 10.1016/j.copsyc.2017.07.012. Epub 2017 Jul 17. PMID 28866434
- [Background] Minassian A, Maihofer AX, Baker DG, Nievergelt CM, Geyer MA, Risbrough VB; Marine Resiliency Study Team. Association of Predeployment Heart Rate Variability With Risk of Postdeployment Posttraumatic Stress Disorder in Active-Duty Marines. JAMA Psychiatry. 2015 Oct;72(10):979-86. doi: 10.1001/jamapsychiatry.2015.0922. PMID 26353072
- [Background] Miranda H, Punnett L, Gore R, Boyer J. Violence at the workplace increases the risk of musculoskeletal pain among nursing home workers. Occup Environ Med. 2011 Jan;68(1):52-7. doi: 10.1136/oem.2009.051474. Epub 2010 Sep 27. PMID 20876554
- [Background] Morgan, J. C., Dill, J., & Kalleberg, A. L. (2013). The quality of healthcare jobs: can intrinsic rewards compensate for low extrinsic rewards? Work, Employment and Society, 27(5), 802-822. doi.org/10.1177/0950017012474707
- [Background] Nam, S., Toneatto, T. The Influence of Attrition in Evaluating the Efficacy and Effectiveness of Mindfulness-Based Interventions. International Journal of Mental Health Addiction 14, 969-981 (2016). https://doi.org/10.1007/s11469-016-9667-1
- [Background] Neff, K. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250. doi.org/10.1080/15298860390209035
- [Background] Neff, K. D. (2020). Commentary on Muris and Otgarr (2020): Let the empirical evidence speak on the self-compassion scale. Min
- [Background] Neff, K. D., Pisitsungkagarn, K., & Hsieh, Y. P. (2008). Self-Compassion and Self- Construal in the United States, Thailand, and Taiwan. Journal of Cross-Cultural Psychology, 39, 267-285. doi.org/10.1177/0022022108314544
- [Background] Neff KD, Toth-Kiraly I, Yarnell LM, Arimitsu K, Castilho P, Ghorbani N, Guo HX, Hirsch JK, Hupfeld J, Hutz CS, Kotsou I, Lee WK, Montero-Marin J, Sirois FM, de Souza LK, Svendsen JL, Wilkinson RB, Mantzios M. Examining the factor structure of the Self-Compassion Scale in 20 diverse samples: Support for use of a total score and six subscale scores. Psychol Assess. 2019 Jan;31(1):27-45. doi: 10.1037/pas0000629. Epub 2018 Aug 20. PMID 30124303
- [Background] O'Brien, W. H., & Carhart, V. (2011). Functional analysis in behavioral medicine settings. European Journal of Psychological Assessment, 27(1), 4-16. doi/10.1027/1015- 5759/a000052
- [Background] O'Brien, W. H., W. H., Horan, K. A., Singh, S., Moeller, M.A., Wasson, R. S., Jex, S. M., Matthews, R. A., & Barratt, C. L. (2017). Preventing Injury, Assault, and Abuse of Nurse Aides Working in Long-Term Residential Settings. Unpublished final technical report for Ohio Occupational Safety and Health Research Program.
- [Background] O'Brien WH, Singh RS, Horan K, Moeller MT, Wasson R, Jex SM. Group-Based Acceptance and Commitment Therapy for Nurses and Nurse Aides Working in Long-Term Care Residential Settings. J Altern Complement Med. 2019 Jul;25(7):753-761. doi: 10.1089/acm.2019.0087. PMID 31314564
- [Background] Petrocchi N, Cheli S. The social brain and heart rate variability: Implications for psychotherapy. Psychol Psychother. 2019 Jun;92(2):208-223. doi: 10.1111/papt.12224. Epub 2019 Mar 20. PMID 30891894
- [Background] Pommier E, Neff KD, Toth-Kiraly I. The Development and Validation of the Compassion Scale. Assessment. 2020 Jan;27(1):21-39. doi: 10.1177/1073191119874108. Epub 2019 Sep 13. PMID 31516024
- [Background] Ramos-Morcillo AJ, Fernandez-Salazar S, Ruzafa-Martinez M, Del-Pino-Casado R. Effectiveness of a Brief, Basic Evidence-Based Practice Course for Clinical Nurses. Worldviews Evid Based Nurs. 2015 Aug;12(4):199-207. doi: 10.1111/wvn.12103. Epub 2015 Jul 28. PMID 26220505
- [Background] Richardson A, Gurung G, Derrett S, Harcombe H. Perspectives on preventing musculoskeletal injuries in nurses: A qualitative study. Nurs Open. 2019 Apr 13;6(3):915-929. doi: 10.1002/nop2.272. eCollection 2019 Jul. PMID 31367415
- [Background] Rolffs JL, Rogge RD, Wilson KG. Disentangling Components of Flexibility via the Hexaflex Model: Development and Validation of the Multidimensional Psychological Flexibility Inventory (MPFI). Assessment. 2018 Jun;25(4):458-482. doi: 10.1177/1073191116645905. Epub 2016 May 5. PMID 27152011
- [Background] Zanchetta MS, Cognet M, Rahman R, Byam A, Carlier P, Foubert C, Lagersie Z, Espindola RF. Blindness, deafness, silence and invisibility that shields racism in nursing education-practice in multicultural hubs of immigration. J Prof Nurs. 2021 Mar-Apr;37(2):467-476. doi: 10.1016/j.profnurs.2020.06.012. Epub 2020 Jul 6. PMID 33867106
- [Background] Schoenfisch AL, Lipscomb HJ. Job characteristics and work organization factors associated with patient-handling injury among nursing personnel. Work. 2009;33(1):117-28. doi: 10.3233/WOR-2009-0847. PMID 19597289
- [Background] Schuster M, Dwyer PA. Post-traumatic stress disorder in nurses: An integrative review. J Clin Nurs. 2020 Aug;29(15-16):2769-2787. doi: 10.1111/jocn.15288. Epub 2020 May 5. PMID 32372541
- [Background] Snyder LA, Chen PY, Vacha-Haase T. The underreporting gap in aggressive incidents from geriatric patients against certified nursing assistants. Violence Vict. 2007;22(3):367-79. doi: 10.1891/088667007780842784. PMID 17619640
- [Background] Snyder CR, Frogner BK, Skillman SM. Facilitating Racial and Ethnic Diversity in the Health Workforce. J Allied Health. 2018 Spring;47(1):58-65. PMID 29504021
- [Background] Spector, P. E., Yang, L. Q., & Zhou, Z. E. (2015). A longitudinal investigation of the role of violence prevention climate in exposure to workplace physical violence and verbal abuse. Work & Stress, 29(4), 325-340. doi.org/10.1080/02678373.2015.1076537
- [Background] Squillace MR, Remsburg RE, Bercovitz A, Rosenoff E, Branden L. An introduction to the National Nursing Assistant Survey. Vital Health Stat 1. 2007 Mar;(44):1-54. PMID 17402361
- [Background] Stanev S, Bailer J, Straker JK, Mehdizadeh S, Park RM, Li H. Worker injuries and safety equipment in Ohio nursing homes. J Gerontol Nurs. 2012 Jun;38(6):47-56. doi: 10.3928/00989134-20120508-01. PMID 22774234
- [Background] Tak S, Sweeney MH, Alterman T, Baron S, Calvert GM. Workplace assaults on nursing assistants in US nursing homes: a multilevel analysis. Am J Public Health. 2010 Oct;100(10):1938-45. doi: 10.2105/AJPH.2009.185421. Epub 2010 Aug 19. PMID 20724680
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Taleghani F, Ashouri E, Saburi M. Empathy, Burnout, Demographic Variables and their Relationships in Oncology Nurses. Iran J Nurs Midwifery Res. 2017 Jan-Feb;22(1):41-45. doi: 10.4103/ijnmr.IJNMR_66_16. PMID 28382057
- [Background] Thayer JF, Ahs F, Fredrikson M, Sollers JJ 3rd, Wager TD. A meta-analysis of heart rate variability and neuroimaging studies: implications for heart rate variability as a marker of stress and health. Neurosci Biobehav Rev. 2012 Feb;36(2):747-56. doi: 10.1016/j.neubiorev.2011.11.009. Epub 2011 Dec 8. PMID 22178086
- [Background] Uthayaratana, T., Taephant, N., & Pisitsungkagarn, K. (2019). Four Noble Truths based problem solving: a therapeutic view. Mental Health, Religion & Culture, 22(2), 119- 129. https://doi.org/10.1080/13674676.2018.1512565
- [Background] Valley MA, Stallones L. Effect of Mindfulness-Based Stress Reduction Training on Health Care Worker Safety: A Randomized Waitlist Controlled Trial. J Occup Environ Med. 2017 Oct;59(10):935-941. doi: 10.1097/JOM.0000000000001090. PMID 28692014
- [Background] Van Gordon, W., & Shonin, E. (2020). Second-Generation Mindfulness-Based Interventions: Toward More Authentic Mindfulness Practice and Teaching. Mindfulness, 11(1). DOI:10.1007/s12671-019-01252-1
- [Background] Wasson RS, Barratt C, O'Brien WH. Effects of Mindfulness-Based Interventions on Self-compassion in Health Care Professionals: a Meta-analysis. Mindfulness (N Y). 2020;11(8):1914-1934. doi: 10.1007/s12671-020-01342-5. Epub 2020 Mar 5. PMID 32421083
- [Background] Wasson, R. S. (2021). Feasibility, Acceptability, and Preliminary Effectiveness of a Pilot Mindful Self-Compassion Intervention for Medical Students. Doctoral Dissertation, Bowling Green State University.
- [Background] Woo T, Ho R, Tang A, Tam W. Global prevalence of burnout symptoms among nurses: A systematic review and meta-analysis. J Psychiatr Res. 2020 Apr;123:9-20. doi: 10.1016/j.jpsychires.2019.12.015. Epub 2020 Jan 22. PMID 32007680
- [Background] White L. Mindfulness in nursing: an evolutionary concept analysis. J Adv Nurs. 2014 Feb;70(2):282-94. doi: 10.1111/jan.12182. Epub 2013 Jun 16. PMID 23772683
- [Background] Whittle R, Mansell G, Jellema P, van der Windt D. Applying causal mediation methods to clinical trial data: What can we learn about why our interventions (don't) work? Eur J Pain. 2017 Apr;21(4):614-622. doi: 10.1002/ejp.964. Epub 2016 Oct 14. PMID 27739626
- [Background] Williams S, Booton T, Watson M, Rowland D, Altini M. Heart Rate Variability is a Moderating Factor in the Workload-Injury Relationship of Competitive CrossFit Athletes. J Sports Sci Med. 2017 Dec 1;16(4):443-449. eCollection 2017 Dec. PMID 29238242
- [Background] Xu, H., O'Brien, W. H., & Chen, Y. (2020). Chinese international student stress and coping: A pilot study of acceptance and commitment therapy. Journal of Contextual Behavioral Science, 15, 135-141. https://doi.org/10.1016/j.jcbs.2019.12.010
- [Background] Young, W., Weckman, G., & Holland, W. (2011). A survey of methodologies for the treatment if missing values within datasets: Limitations and benefit. Theoretical Issues in Ergonomics Science, 12(1),15-43. doi.org/10.1080/14639220903470205
- [Background] Zettle, R. D., Hayes, S. C., Barnes-Holmes, D., & Biglan, A. (2016). The Wiley handbook of contextual behavioral science. John Wiley & Sons.
- [Background] Zhao, J.-B., Ji, J.-L., Yang, X.-L., Yang, Z.-Z., Hou, Y.-F., & Zhang, X.-Y. (2011). National survey of ethical practices among Chinese psychotherapists. Professional Psychology: Research and Practice, 42(5), 375-381. https://doi.org/10.1037/a0025138

DOCUMENTS (1):
  • Informed Consent Form (2024-10-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT06813495/ICF_000.pdf